CLINICAL TRIAL: NCT01253070
Title: A Phase II Study Incorporating Sorafenib (NSC 724772) Into the Therapy of Patients >/= 60 Years of Age With FLT3 Mutated Acute Myeloid Leukemia
Brief Title: Sorafenib Tosylate and Chemotherapy in Treating Older Patients With Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02618; NCI-2011-02618 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000689593; CALGB-11001 (Other: Alliance for Clinical Trials in Oncology); CALGB-11001 (Other: CTEP); U10CA180821 (NIH); U10CA031946 (NIH)
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Results first posted 2016-02-11 (Estimated); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia With FLT3/ITD Mutation; Acute Myeloid Leukemia With Inv(16)(p13.1q22) or t(16;16)(p13.1;q22); CBFB-MYH11; Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; Acute Promyelocytic Leukemia With PML-RARA; FLT3 Gene Mutation; Therapy-Related Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute; Leukemia, Promyelocytic, Acute | interventions — Biopsy; Cytarabine; Daunorubicin; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (daunorubicin, cytarabine, sorafenib tosylate) (Experimental): INDUCTION THERAPY: Daunorubicin hydrochloride 60 mg/m^2/day by IV push or short IV on days 1-3, cytarabine 100 mg/m^2/day by continuous IV on days 1-7, and sorafenib tosylate orally every 12 hours on days 1-7.
  CONSOLIDATION THERAPY - Every 28 days for 2 cycles: Cytarabine 2 g/m^2/day by IV on days 1-5 and sorafenib tosylate 400 mg orally every 12 hours on days 1-28.
  MAINTENANCE - Every 28 days for up to 12 cycles: Sorafenib tosylate 400 mg orally every 12 hours on days 1-28.
  Interventions: Procedure: Biopsy; Procedure: Bone Marrow Aspiration; Drug: Cytarabine; Drug: Daunorubicin Hydrochloride; Other: Laboratory Biomarker Analysis; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Drug: Sorafenib Tosylate

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Bone Marrow Aspiration — Undergo bone marrow aspirate
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-Cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Daunorubicin Hydrochloride — Given IV
  Other Names: Cerubidin; Cerubidine; Cloridrato de Daunorubicina; Daunoblastin; Daunoblastina; Daunoblastine; Daunomycin Hydrochloride; Daunomycin, hydrochloride; Daunorubicin.HCl; Daunorubicini Hydrochloridum; FI-6339; Ondena; RP-13057; Rubidomycin Hydrochloride; Rubilem
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib

SUMMARY:
This phase II trial studies how well sorafenib tosylate and chemotherapy work in treating older patients with acute myeloid leukemia (AML). Sorafenib tosylate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as daunorubicin hydrochloride and cytarabine, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving sorafenib tosylate and combination chemotherapy may be an effective treatment for AML.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if the 1-year overall survival rate of patients age >= 60 with FLT3-ITD AML treated with a sorafenib (sorafenib tosylate) containing induction and post-remission therapy is significantly higher than the historical 1-year overall survival rate of similar patients who were not treated with sorafenib.

SECONDARY OBJECTIVES:

I. To determine the rates of complete remission (CR), CR with incomplete count recovery (CRi), and cytogenetic complete remission (CCyR) to induction chemotherapy.

II. To determine the overall survival, event-free survival, and remission duration in patients treated on this study.

III. To describe the frequency and severity of adverse events for patients treated on this study.

IV. To describe the interaction of pre-treatment disease and patient characteristics including morphology, cytogenetics, immunophenotype, molecular genetic features, white blood cell (WBC) count and hemogram, and performance status on clinical outcomes.

V. To assess FLT3 ligand concentrations and FLT3 plasma inhibitory activity during treatment and determine the relationship to clinical outcomes. (Cancer and Leukemia Group B [CALGB] 21003) VI. To describe the interaction of FLT3 mutation type (tyrosine kinase domain [TKD] vs. ITD) and allelic ratio on clinical outcomes. (CALGB 21003) VII. To characterize geriatric assessment measures in the context of a treatment trial for AML defined by: the observed distribution and number of missing values for each measurement. (CALGB 361006) VIII. To identify specific geriatric assessment measures which are independently associated with overall survival (OS), 30-day treatment-related mortality and key quality of life outcomes (number of days hospitalized, number of oncology clinic visits, admission to a nursing facility) in patients receiving induction chemotherapy for AML. (CALGB 361006) IX. To explore the impact of induction chemotherapy on physical, cognitive, psychosocial factors. (CALGB 361006)

OUTLINE:

INDUCTION THERAPY: Patients receive daunorubicin hydrochloride intravenously (IV) on days 1-3, cytarabine IV continuously on days 1-7, and sorafenib tosylate orally (PO) twice daily (BID) on days 1-7. Patients then undergo a bone marrow aspirate or biopsy on day 14.

Patients with persistent disease undergo a second remission induction therapy comprising daunorubicin hydrochloride IV on days 1-2, cytarabine IV continuously on days 1-5, and sorafenib tosylate PO BID on days 1-7. Patients who achieve complete response (CR)* proceed to consolidation therapy.

CONSOLIDATION THERAPY: Patients** receive cytarabine IV over 3 hours on days 1-5 and sorafenib tosylate PO BID on days 1-28. Treatment repeats every 28 days for 2 cycles in the absence of disease progression or unacceptable toxicity. Patients with continued CR proceed to maintenance therapy.

MAINTENANCE THERAPY: Patients receive sorafenib tosylate PO BID on days 1-28. Treatment repeats every 28 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

NOTE: *Patients who achieve CR and who are eligible for hematopoietic stem cell transplant (HSCT) are encouraged to enroll in Cancer and Leukemia Group B (CALGB) 100103. Patients in CR who are unable or unwilling to undergo HSCT receive two cycles of remission consolidation therapy.

NOTE: ** Patients in CR/complete remission with incomplete count recovery (CRi) who are unable or unwilling to complete remission consolidation therapy may proceed directly to maintenance therapy after consulting with the CALGB study chair.

After completion of study therapy, patients are followed up every 2 months for 2 years, every 3 months for 2 years, and then yearly for a maximum of 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Unequivocal histologic diagnosis of AML according to World Health Organization (WHO) criteria, EXCLUDING:

  * Acute promyelocytic leukemia t(15;17)(q22;q12); promyelocytic leukemia (PML)-retinoic acid receptor, alpha (RARA)
  * Acute myeloid leukemia with t(8;21)(q22;q22); runt-related transcription factor 1 (RUNX1-RUNXT1) as determined by the Ohio State University (OSU) Molecular Reference Laboratory, per CALGB 20202
  * Acute myeloid leukemia with inv(16)(p13.1;q22) or t(16;16(p13.1;q22); core-binding factor, beta subunit (CBFB)-myosin, heavy chain 11, smooth muscle (MYH11) as determined by the OSU Molecular Reference Laboratory, per CALGB 20202
* AML patients with an antecedent hematologic disorder are eligible for treatment on this trial provided that they have not received chemotherapy, including lenalidomide, azacitidine or decitabine for their hematologic disorder; patients with therapy-related AML are eligible if there had been no further exposure to chemotherapy or radiation therapy for > 3 years and their primary malignancy is in remission
* FLT3 mutation (ITD or point mutation) determined by the OSU Molecular Reference Laboratory, per CALGB 20202
* No prior chemotherapy for AML with the following exceptions:

  * Emergency leukapheresis
  * Emergency treatment for hyperleukocytosis with hydroxyurea
  * Cranial radiation therapy (RT) for central nervous system (CNS) leukostasis (one dose only)
  * Growth factor/cytokine support
  * All-trans retinoic acid (ATRA)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2011-04-01 (Actual); Primary Completion 2014-10-31 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey L Uy, Principal Investigator — Alliance for Clinical Trials in Oncology
Locations (43):
- United States (43):
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - AdventHealth Orlando, Orlando, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - Eastern Maine Medical Center, Bangor, Maine
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Christiana Care - Union Hospital, Elkton, Maryland
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Cancer Research Consortium of West Michigan NCORP, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Spectrum Health Reed City Hospital, Reed City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Northwell Health NCORP, Lake Success, New York
  - Northwell Health/Center for Advanced Medicine, Lake Success, New York
  - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - NYP/Weill Cornell Medical Center, New York, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Vidant Oncology-Kinston, Kinston, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Cancer Care Associates-Norman, Norman, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Roper Hospital, Charleston, South Carolina
  - Central Vermont Medical Center/National Life Cancer Treatment, Berlin Corners, Vermont
  - University of Vermont and State Agricultural College, Burlington, Vermont
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

REFERENCES:
- [Derived] Seffernick AE, Mrozek K, Nicolet D, Stone RM, Eisfeld AK, Byrd JC, Archer KJ. High-dimensional genomic feature selection with the ordered stereotype logit model. Brief Bioinform. 2022 Nov 19;23(6):bbac414. doi: 10.1093/bib/bbac414. PMID 36184192
- [Derived] Mims AS, Kohlschmidt J, Borate U, Blachly JS, Orwick S, Eisfeld AK, Papaioannou D, Nicolet D, Mromicronzek K, Stein E, Bhatnagar B, Stone RM, Kolitz JE, Wang ES, Powell BL, Burd A, Levine RL, Druker BJ, Bloomfield CD, Byrd JC. A precision medicine classification for treatment of acute myeloid leukemia in older patients. J Hematol Oncol. 2021 Jun 23;14(1):96. doi: 10.1186/s13045-021-01110-5. PMID 34162404
- [Derived] Klepin HD, Ritchie E, Major-Elechi B, Le-Rademacher J, Seisler D, Storrick L, Sanford BL, Marcucci G, Zhao W, Geyer SA, Ballman KV, Powell BL, Baer MR, Stock W, Cohen HJ, Stone RM, Larson RA, Uy GL. Geriatric assessment among older adults receiving intensive therapy for acute myeloid leukemia: Report of CALGB 361006 (Alliance). J Geriatr Oncol. 2020 Jan;11(1):107-113. doi: 10.1016/j.jgo.2019.10.002. Epub 2019 Oct 24. PMID 31668825
- [Derived] Yin J, LaPlant B, Uy GL, Marcucci G, Blum W, Larson RA, Stone RM, Mandrekar SJ. Evaluation of event-free survival as a robust end point in untreated acute myeloid leukemia (Alliance A151614). Blood Adv. 2019 Jun 11;3(11):1714-1721. doi: 10.1182/bloodadvances.2018026112. PMID 31171508
- [Derived] Uy GL, Mandrekar SJ, Laumann K, Marcucci G, Zhao W, Levis MJ, Klepin HD, Baer MR, Powell BL, Westervelt P, DeAngelo DJ, Stock W, Sanford B, Blum WG, Bloomfield CD, Stone RM, Larson RA. A phase 2 study incorporating sorafenib into the chemotherapy for older adults with FLT3-mutated acute myeloid leukemia: CALGB 11001. Blood Adv. 2017 Jan 24;1(5):331-340. doi: 10.1182/bloodadvances.2016003053. PMID 29034366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 54 participants were recruited from April 2011 to August 2013.
Groups:
- Treatment (Daunorubicin, Cytarabine, Sorafenib Tosylate): INDUCTION THERAPY: Daunorubicin hydrochloride 60 mg/m^2/day by IV push or short IV on days 1-3, cytarabine 100 mg/m^2/day by continuous IV on days 1-7, and sorafenib tosylate 400 mg orally every 12 hours on days 1-7.
  CONSOLIDATION THERAPY - Every 28 days for 2 cycles: Cytarabine 2 g/m^2/day by IV on days 1-5 and sorafenib tosylate 400 mg orally every 12 hours on days 1-28.
  MAINTENANCE - Every 28 days for up to 12 cycles: Sorafenib tosylate 400 mg orally every 12 hours on days 1-28.
Period: Overall Study
Arm/Group | Treatment (Daunorubicin, Cytarabine, Sorafenib Tosylate)
Started | 54
Completed | 54
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Daunorubicin, Cytarabine, Sorafenib Tosylate)
Number analyzed (Participants) | 54
Age, Continuous [Median (Full Range); unit: years] | 67.4 [60.3 to 82.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 51
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 54
FLT3 Mutation [Number; unit: participants] — FLT3 (FMS-like tyrosine kinase-3) mutation testing at baseline was performed centrally for all patients. Participants were eligible for the study if they had an ITD (internal tandem duplication) or TKD (tyrosine kinase domain) mutation.
  participants
    ITD | 39
    TKD | 15

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Rate
Description: Percentage of patients who were alive at 1 year. The analysis was split between patients with having a FLT3 (FMS-like tyrosine kinase-3) ITD (internal tandem duplication) or TKD (tyrosine kinase domain) mutation. The FLT3 mutation testing at baseline was performed centrally for all patients.
Time Frame: 1 year
Population: Three participants withdrew consent to protocol treatment and follow-up prior to 1 year post registration (2 ITD; 1 TKD). These participants have been excluded from the primary endpoint analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- ITD Mutated Participants; TKD Mutated Participants: INDUCTION THERAPY: Daunorubicin hydrochloride 60 mg/m^2/day by IV push or short IV on days 1-3, cytarabine 100 mg/m^2/day by continuous IV on days 1-7, and sorafenib tosylate 400 mg orally every 12 hours on days 1-7.
  CONSOLIDATION THERAPY - Every 28 days for 2 cycles: Cytarabine 2 g/m^2/day by IV on days 1-5 and sorafenib tosylate 400 mg orally every 12 hours on days 1-28.
  MAINTENANCE - Every 28 days for up to 12 cycles: Sorafenib tosylate 400 mg orally every 12 hours on days 1-28.
Arm/Group | ITD Mutated Participants | TKD Mutated Participants
Number analyzed (Participants) | 37 | 14
percentage of participants | 62 [45 to 78] | 71 [42 to 92]

2. Secondary Outcome: OS
Description: OS was defined as the time from registration to death of any cause. Surviving patients were censored at the date of last follow-up. The median OS with 95% confidence interval (CI) was estimated using the Kaplan Meier method.
Time Frame: Time from registration to death (up to 10 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ITD Mutated Participants | TKD Mutated Participants
Number analyzed (Participants) | 39 | 15
months | 15 [10.4 to 20.1] | 16.2 [5.0 to NA] — The upper limit was not calculable because an insufficient number of participants reached the event at the final time point for assessment

3. Secondary Outcome: Event-free Survival
Description: Event-free survival (EFS) was defined as the time for registration to failure to achieve CR during induction, relapse or death. Participants without events were censored at date of last follow-up. The median EFS with 95% CI was estimated using the Kaplan Meier method.
Time Frame: Time from registration to death or relapse (up to 10 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ITD Mutated Participants | TKD Mutated Participants
Number analyzed (Participants) | 39 | 15
months | 8.8 [3.0 to 13.9] | 7.8 [1.3 to 11.6]

ADVERSE EVENTS:
Description: At the time of analysis, adverse event data was collected on 50 of 54 participants.
Arm/Group | Treatment (Daunorubicin, Cytarabine, Sorafenib Tosylate)
Serious Adverse Events (participants affected / at risk) | 21/50
Other Adverse Events (participants affected / at risk) | 42/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Daunorubicin, Cytarabine, Sorafenib Tosylate) (N=50)
Anemia (Blood and lymphatic system disorders) | 20 (24)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 (2)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 13 (15)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 5 (5)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrioventricular block first degree (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2)
Cardiac disorders - Other (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Heart failure (Cardiac disorders) | 2 (2)
Left ventricular systolic dysfunction (Cardiac disorders) | 3 (3)
Pericarditis (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 4 (4)
Supraventricular tachycardia (Cardiac disorders) | 2 (2)
Ventricular arrhythmia (Cardiac disorders) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Blurred vision (Eye disorders) | 2 (2)
Dry eye (Eye disorders) | 1 (1)
Eye disorders - Other (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Constipation (Gastrointestinal disorders) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 14 (14)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 7 (9)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (5)
Chills (General disorders) | 1 (1)
Edema limbs (General disorders) | 7 (9)
Fatigue (General disorders) | 11 (13)
Fever (General disorders) | 1 (1)
Localized edema (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 2 (7)
Allergic reaction (Immune system disorders) | 1 (2)
Bone infection (Infections and infestations) | 1 (2)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Infections and infestations - Other (Infections and infestations) | 1 (1)
Laryngitis (Infections and infestations) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 8 (10)
Sepsis (Infections and infestations) | 6 (7)
Urinary tract infection (Infections and infestations) | 4 (4)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 3 (3)
Alanine aminotransferase increased (Investigations) | 8 (8)
Alkaline phosphatase increased (Investigations) | 6 (7)
Aspartate aminotransferase increased (Investigations) | 11 (11)
Blood bilirubin increased (Investigations) | 8 (8)
Creatinine increased (Investigations) | 5 (5)
Ejection fraction decreased (Investigations) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
INR increased (Investigations) | 4 (6)
Investigations - Other (Investigations) | 2 (4)
Lymphocyte count decreased (Investigations) | 8 (10)
Neutrophil count decreased (Investigations) | 19 (22)
Platelet count decreased (Investigations) | 20 (23)
Urine output decreased (Investigations) | 1 (1)
Weight gain (Investigations) | 1 (1)
Weight loss (Investigations) | 2 (2)
White blood cell decreased (Investigations) | 14 (15)
Acidosis (Metabolism and nutrition disorders) | 3 (3)
Alkalosis (Metabolism and nutrition disorders) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (9)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 11 (11)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 13 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 11 (11)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 10 (10)
Hypomagnesemia (Metabolism and nutrition disorders) | 5 (5)
Hyponatremia (Metabolism and nutrition disorders) | 11 (13)
Hypophosphatemia (Metabolism and nutrition disorders) | 8 (11)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 5 (5)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 (2)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysarthria (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Lethargy (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Reversible posterior leukoencephalopathy syndrome (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Confusion (Psychiatric disorders) | 4 (4)
Insomnia (Psychiatric disorders) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Chronic kidney disease (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 2 (2)
Renal calculi (Renal and urinary disorders) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 (13)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (3)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (4)
Hypotension (Vascular disorders) | 5 (6)
Thromboembolic event (Vascular disorders) | 2 (3)
Vascular disorders - Other (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Daunorubicin, Cytarabine, Sorafenib Tosylate) (N=50)
Anemia (Blood and lymphatic system disorders) | 41 (134)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 1 (7)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 5 (6)
Febrile neutropenia (Blood and lymphatic system disorders) | 27 (37)
Lymph node pain (Blood and lymphatic system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 3 (8)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Mitral valve disease (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 6 (7)
Sinus tachycardia (Cardiac disorders) | 2 (3)
Ventricular arrhythmia (Cardiac disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 3 (3)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 3 (3)
Blurred vision (Eye disorders) | 4 (5)
Conjunctivitis (Eye disorders) | 2 (4)
Dry eye (Eye disorders) | 1 (1)
Eye disorders - Other (Eye disorders) | 2 (2)
Vitreous hemorrhage (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 13 (18)
Anal ulcer (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 20 (25)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 35 (81)
Dry mouth (Gastrointestinal disorders) | 4 (6)
Dyspepsia (Gastrointestinal disorders) | 4 (5)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 4 (8)
Gastritis (Gastrointestinal disorders) | 2 (4)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 5 (7)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 2 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 (2)
Hemorrhoids (Gastrointestinal disorders) | 6 (7)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 22 (31)
Nausea (Gastrointestinal disorders) | 30 (58)
Oral hemorrhage (Gastrointestinal disorders) | 3 (3)
Oral pain (Gastrointestinal disorders) | 4 (5)
Rectal pain (Gastrointestinal disorders) | 2 (3)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 12 (18)
Chills (General disorders) | 12 (14)
Edema face (General disorders) | 3 (3)
Edema limbs (General disorders) | 22 (37)
Facial pain (General disorders) | 1 (1)
Fatigue (General disorders) | 31 (77)
Fever (General disorders) | 12 (14)
General disorders and administration site conditions - Other (General disorders) | 2 (4)
Infusion related reaction (General disorders) | 2 (2)
Malaise (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 8 (11)
Hepatobiliary disorders - Other (Hepatobiliary disorders) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1)
Bone infection (Infections and infestations) | 1 (2)
Catheter related infection (Infections and infestations) | 5 (5)
Infections and infestations - Other (Infections and infestations) | 8 (9)
Lip infection (Infections and infestations) | 2 (2)
Lung infection (Infections and infestations) | 3 (5)
Pharyngitis (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 3 (3)
Sinusitis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 2 (2)
Small intestine infection (Infections and infestations) | 1 (2)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 5 (6)
Bruising (Injury, poisoning and procedural complications) | 7 (7)
Fall (Injury, poisoning and procedural complications) | 4 (4)
Activated partial thromboplastin time prolonged (Investigations) | 7 (10)
Alanine aminotransferase increased (Investigations) | 26 (66)
Alkaline phosphatase increased (Investigations) | 17 (28)
Aspartate aminotransferase increased (Investigations) | 23 (52)
Blood bilirubin increased (Investigations) | 25 (49)
Cholesterol high (Investigations) | 2 (2)
Creatinine increased (Investigations) | 9 (19)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
INR increased (Investigations) | 11 (22)
Investigations - Other (Investigations) | 2 (4)
Lipase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 21 (68)
Neutrophil count decreased (Investigations) | 42 (97)
Platelet count decreased (Investigations) | 42 (133)
Serum amylase increased (Investigations) | 1 (1)
Weight loss (Investigations) | 7 (11)
White blood cell decreased (Investigations) | 30 (71)
Anorexia (Metabolism and nutrition disorders) | 22 (38)
Dehydration (Metabolism and nutrition disorders) | 3 (6)
Hypercalcemia (Metabolism and nutrition disorders) | 4 (8)
Hyperglycemia (Metabolism and nutrition disorders) | 27 (69)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (5)
Hypermagnesemia (Metabolism and nutrition disorders) | 6 (6)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 3 (3)
Hyperuricemia (Metabolism and nutrition disorders) | 2 (3)
Hypoalbuminemia (Metabolism and nutrition disorders) | 34 (67)
Hypocalcemia (Metabolism and nutrition disorders) | 24 (36)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 24 (37)
Hypomagnesemia (Metabolism and nutrition disorders) | 12 (20)
Hyponatremia (Metabolism and nutrition disorders) | 24 (40)
Hypophosphatemia (Metabolism and nutrition disorders) | 22 (31)
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 3 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (15)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 7 (8)
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness right-sided (Musculoskeletal and connective tissue disorders) | 2 (2)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (6)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Dizziness (Nervous system disorders) | 12 (15)
Dysgeusia (Nervous system disorders) | 3 (3)
Headache (Nervous system disorders) | 16 (20)
Lethargy (Nervous system disorders) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (1)
Nervous system disorders - Other (Nervous system disorders) | 2 (2)
Neuralgia (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (12)
Phantom pain (Nervous system disorders) | 1 (1)
Sinus pain (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Transient ischemic attacks (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 2 (2)
Anxiety (Psychiatric disorders) | 9 (10)
Confusion (Psychiatric disorders) | 3 (3)
Depression (Psychiatric disorders) | 6 (6)
Hallucinations (Psychiatric disorders) | 2 (2)
Insomnia (Psychiatric disorders) | 9 (14)
Personality change (Psychiatric disorders) | 1 (2)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 4 (9)
Proteinuria (Renal and urinary disorders) | 3 (8)
Renal and urinary disorders - Other (Renal and urinary disorders) | 3 (10)
Urinary frequency (Renal and urinary disorders) | 5 (9)
Urinary incontinence (Renal and urinary disorders) | 2 (2)
Vaginal hemorrhage (Reproductive system and breast disorders) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 13 (21)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 18 (25)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 (14)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Pharyngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 (9)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 8 (12)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 3 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (19)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4 (5)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (5)
Pain of skin (Skin and subcutaneous tissue disorders) | 2 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 9 (18)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (10)
Purpura (Skin and subcutaneous tissue disorders) | 3 (3)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 30 (63)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 11 (26)
Skin ulceration (Skin and subcutaneous tissue disorders) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Flushing (Vascular disorders) | 1 (1)
Hematoma (Vascular disorders) | 1 (1)
Hot flashes (Vascular disorders) | 2 (5)
Hypertension (Vascular disorders) | 17 (30)
Hypotension (Vascular disorders) | 11 (13)
Phlebitis (Vascular disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (2)
Vascular disorders - Other (Vascular disorders) | 1 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less